CLINICAL TRIAL: NCT02445911
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of KQ-791 in Subjects With Type 2 Diabetes
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of KQ-791 in Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaneq Bioscience Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KQ-791-02
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- KQ-791 Dose 1 (Experimental): Single loading dose on day 1, followed by single doses on days 8, 15, 22, 29
  Interventions: Drug: KQ-791
- KQ-791 Dose 2 (Experimental): Single loading dose on day 1, followed by a daily dose for 28 days
  Interventions: Drug: KQ-791
- KQ-791 Dose 3 (Experimental): Single loading dose on day 1 or days 1-2, followed by a daily dose for 28 days
  Interventions: Drug: KQ-791
- Placebo (Placebo Comparator): Multiple ascending doses matching KQ-791 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KQ-791 — Capsules administered orally
  Arms: KQ-791 Dose 1; KQ-791 Dose 2; KQ-791 Dose 3
Drug: Placebo — Capsules administered orally
  Arms: Placebo

SUMMARY:
This study will consist of multiple ascending oral doses in up to 3 groups, for 29 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type 2 Diabetes Mellitus (T2DM)
* Be an adult between the ages of 18 (19 for Lincoln site) and 70 years
* Female participants must be of non-childbearing potential, and must be either 1) postmenopausal with amenorrhea for at least 1 year prior to the first dose and Follicle Stimulating Hormone (FSH) serum levels consistent with postmenopausal status, or 2) have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

  * hysteroscopic sterilization
  * bilateral tubal ligation or bilateral salpingectomy
  * hysterectomy
  * bilateral oophorectomy
* Non-vasectomized males must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 100 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dosing. A male who has been vasectomized less than 4 months prior to first dosing must follow the same restrictions as a non-vasectomized male)
* Males must agree to not donate sperm during the study and for 100 days following the last dose
* Have an HbA1c value between 7.0-10.0%
* Be on a stable treatment regimen of metformin, with or without diet/exercise, for at least 8 weeks
* Weigh 60 kilograms (kg) or more at screening and have a body mass index (BMI) greater than or equal to (≥) 25.0 and less than or equal to (≤) 40.0 kilograms/meters squared (kg/m2)
* Have laboratory test results within the normal range for T2DM population, or with abnormalities deemed clinically insignificant. Urine protein levels must be within normal limits
* Absence of active diabetic retinopathy (Stage 2 or greater by the International Clinical Disease Severity Scale for Diabetic Retinopathy)
* Are willing to comply with specific dietary restrictions (that is, [i] able to fast overnight for at least 8-12 hours on several days and [ii] able to consume the standard meals provided during specified confinement days)
* Have given written consent to allow collection of samples for Peripheral Blood Mononuclear Cells (PBMC) analysis and for possible biomarkers/safety analysis
* Have given written informed consent approved by the institutional review board (IRB) governing the site

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Participated (defined as the last dose of study drug) within 30 days prior to dosing in a clinical trial involving an investigational product or non-approved use of a drug with a short half-life or within 5 half-lives of an investigational product with a half-life longer than 6 days
* - Have a (QTcF) greater than (>) 450 milliseconds (msec), or clinical significant hypokalemia, a family history of long QT syndrome or any abnormality in the 12-lead Electrocardiogram (ECG)
* Abnormal blood pressure (sitting) defined as diastolic blood pressure > 95 or less than (<) 50 millimeter of mercury (mmHg) and/or systolic blood pressure > 160 or < 90 mmHg
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Show evidence of regular use of known drugs of abuse and/or positive findings on urinary drug screening
* Evidence of human immunodeficiency virus (HIV) infection, hepatitis B, hepatitis C and/or positive results at screening for the respective antibodies for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV)
* Have anemia that would interfere with the trial or have donated ≥500 mL of blood within 56 days before the first dose or have donated plasma within 7 days before the first dose or provided any blood donation within last 30 days
* Have an average weekly alcohol intake that exceeds 14 units per week (males) and 7 units per week (females) [1 unit = 12 ounces (oz) or 360 mL of beer, 5 oz or 150 mL of wine, or 1.5 oz or 45 mL of distilled spirits] or are unwilling to stop alcohol consumption 48 hours prior to the first dosing and throughout the study
* Consume more than 10 cigarettes per day or the equivalent or are unable or unwilling to adhere to restricted smoking policies
* Have had >1 episode of documented severe hypoglycemia within last 6 months or are currently diagnosed as having hypoglycemia unawareness
* Have any of the following clinical laboratory test results:

  * estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (impaired renal function)
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 1.5 times (x) the upper limit of normal (ULN)
  * triglycerides (TG) > 500 milligrams/deciliter (mg/dL)
* Have used insulin or other glycemic control medications, except metformin, for diabetic control within 3 months
* Intend to use non-steroidal anti-inflammatory drugs (except aspirin) and drugs known to prolong QT interval, herbal products, or vitamin supplements that change glucose levels. The following medications are allowed for participants:

  * drugs for treatment of hypertension or lipid disorders (except bile acid resins, niacin or fish oils), platelet inhibitors, and on stable dose for 12 weeks prior to first dose
  * thyroid replacement therapy, proton pump inhibitors, antidepressants, antihistamines, regularly taken over-the-counter (OTC) and anti-emetics that do not cause a corrected QT interval (QTc) prolongation, provided such drugs are not specifically excluded
  * hormonal replacement therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email: daniel.bouthillier@Kaneq.ca, Study Director — Kaneq Bioscience
Locations (4):
- United States (4):
  - Celerion, Tempe, Arizona
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Celerion, Lincoln, Nebraska

RESULTS

PARTICIPANT FLOW:
Groups:
- KQ-791 Dose 1: Single loading dose of 100 mg on day 1, followed by single 50 mg doses on days 8, 15, 22, 29
  KQ-791: Capsules administered orally
- KQ-791 Dose 2: Single loading dose of 250 mg on day 1, followed by a daily dose of 25 mg for 28 days
  KQ-791: Capsules administered orally
- KQ-791 Dose 3: Single loading dose of 1500 mg on day 1, followed by a daily dose of 150 mg for 28 days
  KQ-791: Capsules administered orally
Period: Overall Study
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Started | 20 | 20 | 21 | 20
Completed | 20 | 20 | 21 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 20 | 16 | 67
  >=65 years | 3 | 6 | 1 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 10 | 10 | 42
  Male | 8 | 10 | 11 | 10 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 19 | 17 | 16 | 69
  Not Hispanic or Latino | 3 | 1 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 2 | 5 | 12
  White | 17 | 18 | 19 | 15 | 69
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 21 | 20 | 81

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Change From Baseline in Fasting Blood Glucose Between KQ-791 and Placebo
Description: Data table is change from baseline in Fasting Blood Glucose. Statistical Analysis includes results for difference in Change from baseline in Fasting Blood Glucose Between KQ-791 and Placebo.
Time Frame: Baseline to Day 29
Population: Pharmacodynamic (PD) population incudes all 81 participants
Measure: Mean (Standard Deviation); unit: mg/dL milligrams per deciliters
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
mg/dL milligrams per deciliters | -3.28 (22.99) | -3.93 (30.63) | 0.67 (30.82) | 3.17 (23.17)
Statistical Analysis 1: Comparison: KQ-791 Dose 1 vs Placebo; Test type: Other; Least-squares Mean Difference = -6.78, 95% CI 2-sided [-23.75 to 10.18] — Least-squares means have baseline and site as covariates. Placebo was the reference group
Statistical Analysis 2: Comparison: KQ-791 Dose 2 vs Placebo; Test type: Other; Least-squares Mean Difference = -2.97, 95% CI 2-sided [-19.65 to 13.72] — Least-squares means have baseline and site as covariates. Placebo was the reference group
Statistical Analysis 3: Comparison: KQ-791 Dose 3 vs Placebo; Test type: Other; Least-squares Mean Difference = -5.05, 95% CI 2-sided [-21.97 to 11.88] — Least-squares means have baseline and site as covariates. Placebo was the reference group

2. Primary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Events
Time Frame: Baseline to Day 29
Population: PD population includes all 81 participants
Measure: Number; unit: participants
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
participants | 12 | 12 | 11 | 14

3. Secondary Outcome: Change From Baseline in the Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: QUICKI = 1/(log FPG + log FPI) where FPG = fasting plasma glucose (mg/dL); FPI = fasting plasma insulin (estimated based on fasting serum insulin; (μIU/mL)). Lower numbers reflect greater insulin resistance.
Time Frame: Baseline to Day 29
Population: PD population includes all 81 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
units on a scale | .0043 (.012) | .003 (.013) | .005 (.0125) | -.0012 (.0116)

4. Secondary Outcome: Change From Baseline in the Insulin Sensitivity Index (ISI)
Description: Insulin sensitivity index (ISI) composite using Matsuda's whole body insulin sensitivity, ISI [composite] = 10000/√[(FPG x FPI)x(Mean Glucose 0-120min in MMTT x Mean Insulin 0-120 min in MMTT)] where MMTT is a mixed meal tolerance test, Hour 0=just prior dosing. Lower values indicate greater insulin resistance.
Time Frame: Baseline to Day 29
Population: Includes all subjects who receive at least one dose of study drug and have evaluable ISI data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 19 | 21 | 20
units on a scale | .0043 (0.7345) | -.0585 (0.586) | 0.145 (0.697) | -0.112 (0.669)

5. Secondary Outcome: Change From Baseline in Beta Cell Function
Description: Evaluated as beta index = (Insulin Area Under the Effect Curve (AUEC) in MMTT/Glucose AUEC in MMTT)
Time Frame: Baseline to Day 29
Population: PD population includes all 81 participants
Measure: Mean (Standard Deviation); unit: (hr*μIU/mL(hr*mg/dL))
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
(hr*μIU/mL(hr*mg/dL)) | 0.00098 (0.0866) | 0.012 (0.0585) | 0.0535 (0.1099) | 0.0027 (0.0491)

6. Secondary Outcome: Change From Baseline in Disposition Index
Description: Disposition Index evaluated as beta index x ISI [composite]. Lower values of the disposition index suggests loss of function of beta cells.
Time Frame: Baseline to Day 29
Population: Includes all subjects who receive at least one dose of study drug and have evaluable data for disposition index.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 19 | 21 | 20
Index | 0.022 (0.128) | 0.023 (0.147) | 0.084 (0.185) | 0.008 (0.085)

7. Secondary Outcome: Change From Baseline in the Hepatic Insulin Resistance Index
Description: Hepatic Insulin Resistance Index will be evaluated as Glucose AUEC from zero to 30 minutes (AUEC0-30min) in MMTT x Insulin AUEC0-30 min in MMTT
Time Frame: Baseline to Day 29
Population: PD population includes all 81 participants
Measure: Mean (Standard Deviation); unit: (hr*mg/dL)*(hr*μUI/mL)
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
(hr*mg/dL)*(hr*μUI/mL) | 99.51 (495.81) | 255.53 (484.27) | 93.17 (462.25) | 56.90 (482.72)

8. Secondary Outcome: Change From Baseline in 7-point Average Blood Glucose
Description: The 7-points measured were just prior to each meal and 90 minutes after the start of the meal and approximately bedtime.
Time Frame: Baseline to Day 29
Population: PD population includes all 81 participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
mg/dL | -5.04 (20.76) | 0.35 (35.74) | -2.61 (38.66) | 4.44 (27.91)

9. Secondary Outcome: Change From Baseline in Postprandial Glucose
Time Frame: Baseline to Day 29
Population: PD population includes all 81 participants
Measure: Mean (Standard Deviation); unit: hr*mg/dL
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 20
hr*mg/dL | -72.23 (281.62) | -0.086 (484.712) | -35.60 (524.57) | 58.61 (381.88)

10. Secondary Outcome: Change From Baseline in HbA1c
Time Frame: Baseline to Day 29
Population: Includes all subjects who receive at least one dose of study drug and have evaluable HbA1c data.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 18
Percentage of glycosylated hemoglobin | -0.185 (0.3265) | 0.025 (0.4303) | -0.315 (0.5174) | -0.0333 (0.3343)

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24-hours Post-Dose (AUC0-24)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AUC0-24.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
ng*hr/mL | 14372.2 (2882.69) | 29011.2 (6030.57) | 140990.4 (47460.96)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
ng/mL | 747.56 (163.768) | 1484.74 (341.712) | 7204.70 (2517.201)

13. Secondary Outcome: Time of the Maximum Measured Plasma Concentration (Tmax)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Tmax.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
hours | 4.60 (3.251) | 5.05 (3.395) | 9.42 (8.663)

14. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUCtau)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose; Day 3, 8, 15, 22, 29, and up to 24 hours post-dose on Day 29
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AUCtau.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
ng*hr/mL | 76863.5 (34469.47) | 25754.9 (13130.00) | 150681.0 (55372.30)

15. Secondary Outcome: Maximum Observed Plasma Concentration at Steady-state (Cmax_ss)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose; Day 3, 8, 15, 22, 29, and up to 24 hours post-dose on Day 29
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Cmax_ss.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
ng/mL | 657.82 (238.542) | 1164.65 (568.489) | 7221.37 (2672.180)

16. Secondary Outcome: Time of the Maximum Measured Plasma Concentration at Steady-state (Tmax_ss)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose; Day 3, 8, 15, 22, 29, and up to 24 hours post-dose on Day 29
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute Tmax_ss.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
hours | 5.10 (5.00) | 5.43 (5.69) | 3.83 (3.40)

17. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose; Day 3, 8, 15, 22, 29, and up to 24 hours post-dose on Day 29
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute t1/2.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 20 | 20 | 21
hours | 201.095 (79.378) | 184.386 (36.385) | 178.018 (28.389)

18. Secondary Outcome: Accumulation Index (AI)
Description: Based on AUC (RacAUC), where RacAUC is the ratio of AUC during a dosing interval following the last dose over the loading dose (first dose)
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose; Day 3, 8, 15, 22, 29, and up to 24 hours post-dose on Day 29
Population: Includes all randomized subjects who received at least 1 dose of KQ-791and had sufficient evaluable PK data to compute AI.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3
Number analyzed (Participants) | 19 | 20 | 21
1/h | 1.97 (0.537) | 9.37 (4.934) | 12.01 (6.507)

ADVERSE EVENTS:
Arm/Group | KQ-791 Dose 1 | KQ-791 Dose 2 | KQ-791 Dose 3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 1/20
Other Adverse Events (participants affected / at risk) | 12/20 | 12/20 | 11/21 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KQ-791 Dose 1 (N=20) | KQ-791 Dose 2 (N=20) | KQ-791 Dose 3 (N=21) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KQ-791 Dose 1 (N=20) | KQ-791 Dose 2 (N=20) | KQ-791 Dose 3 (N=21) | Placebo (N=20)
Conjunctival irritation (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 2 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 3 | 5 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0
Glomuerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 7 | 5 | 6 | 4
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written consent